CLINICAL TRIAL: NCT02248675
Title: An Adjunctive Behavioral Sleep Intervention to Prevent Veteran Suicides
Brief Title: Adjunctive Brief Behavioral Treatment of Insomnia (BBTI) for Sleep Intervention (SI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: PPO 13-373; I21HX001473 (NIH)
Record Dates: First submitted 2014-09-22; First posted 2014-09-25 (Estimated); Results first posted 2017-04-28 (Actual); Last update posted 2017-04-28 (Actual); Status verified 2017-03

CONDITIONS: Insomnia; Depression; Posttraumatic Stress Disorder; Suicidal Ideation
Keywords: sleep disorders; insomnia; suicidal ideation; Depression; Depressive disorders; PTSD; anxiety disorders; suicide; cognitive behavioral therapy
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Depression; Stress Disorders, Post-Traumatic; Suicidal Ideation; Sleep Wake Disorders; Depressive Disorder; Anxiety Disorders; Suicide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CBT-I + TAU (Experimental): Cognitive Behavioral Therapy for Insomnia (CBT-I), an evidence-based insomnia treatment. In this study it will be delivered in four individual sessions as an adjunctive treatment to treatment as usual (TAU).
  Interventions: Behavioral: CBT-I; Other: TAU
- TAU (Active Comparator): Treatment as Usual: All participants will be encouraged to begin or continue treatment of co-occurring conditions as recommended by treatment providers. This may include treatment within the primary care teams, through behavioral telehealth, and/or specialty outpatient mental health. Participants randomized to TAU may receive pharmacotherapy for insomnia, though CBT-I will be precluded until after the post-treatment assessments.
  Interventions: Other: TAU

INTERVENTIONS:
Behavioral: CBT-I — Cognitive Behavioral Therapy for Insomnia (CBT-I), an evidence-based insomnia treatment. In this study it will be delivered in four individual sessions.
  Arms: CBT-I + TAU
Other: TAU — Treatment as Usual: All participants will be encouraged to begin or continue treatment of co-occurring conditions as recommended by treatment providers. This may include treatment within the primary care teams, through behavioral telehealth, and/or specialty outpatient mental health. Participants randomized to TAU may receive pharmacotherapy for insomnia, though CBT-I will be precluded until after the post-treatment assessments.

SUMMARY:
There is a strong association between sleep disturbance and suicidal thoughts and behaviors. Sleep disturbance is also highly comorbid with other common conditions associated with suicide such as depression and posttraumatic stress disorder. Accordingly, this application focuses on improving sleep as a novel suicide prevention strategy that can be delivered to a broad range of Veterans. This pilot proposal specifically examines how Cognitive Behavioral Therapy for Insomnia, an efficacious treatment for insomnia, may reduce suicidal ideation in Veterans who also suffer from additional conditions. The proposal further suggests that adding this sleep intervention to usual care may further enhance overall care by increasing the utilization of recommended treatments for depression and posttraumatic stress disorder.

DETAILED DESCRIPTION:
Anticipated Benefit to VA Healthcare The proposed study will establish proof of concept that suicidal ideation can be reduced by adjunctively treating insomnia, a common problem that is both a risk factor for suicide and highly prevalent in common conditions associated with suicide such as depression and PTSD. In addition, to the extent that insomnia is improved, the investigators expect to both enhance Veteran's quality of life and increase their engagement with treatments for co-occurring conditions.

Project Background Suicide is the tenth leading cause of death in the U.S., is a major concern of the Department of Veterans Affairs (VA), and occurs at elevated rates among Veterans. Veterans with common chronic conditions such as PTSD, depression, substance abuse and chronic pain are at increased risk for suicide. Although evidence-based treatments exist for these conditions, a significant number of Veterans do not engage in or complete such treatments. This application focuses on an intervention target that co-occurs in each of the listed conditions at high rates and is itself an independent risk factor for suicidal thoughts and behaviors: the sleep disturbance of insomnia. Therefore, this proposal examines the use of cognitive-behavioral therapy for insomnia (CBT-I), an efficacious intervention that targets insomnia, as a novel way to reduce suicidal ideation in at-risk Veterans. Importantly, CBT-I has been successfully used in patients with PTSD and depression. Preliminary evidence from an uncontrolled trial in civilians suggests that CBT-I may also decrease suicidal ideation, but this has not been tested in Veterans, in the context of treatments for co-occurring conditions, or in a controlled trial.

Project Objectives The ultimate goal of the broader program of research is to reduce suicide among Veterans, while the proposed pilot project will provide data to guide the development of a larger trial. The primary objectives of this pilot project are to test whether using CBT-I as an adjunctive treatment: (1) is feasible to deliver in the context of other ongoing care and acceptable to participants; (2) can reduce the severity of suicidal ideation among Veterans at risk for suicide; and (3) can increase rates of engagement in treatments that address the co-morbid conditions that also put them at risk for suicide. The latter objective will help refine the study methods, design, and intervention in anticipation of a larger trial.

Project Methods In order to achieve these proof-of-concept objectives the investigators will conduct a small randomized clinical trial. Veterans who are either flagged as high risk for suicide or who have depression or PTSD will be recruited from VA sites only. Approximately 56 such Veterans who also endorse current suicidal ideation and current insomnia will be randomized to receive either treatment-as-usual or a 4-session CBT-I treatment in addition to treatment-as-usual. All participants will be encouraged to continue or to seek treatment for co-occurring conditions as recommended by their VA treatment providers. Assessments of suicidal ideation, insomnia, depression, PTSD, and quality of life will be conducted at baseline and following the treatment period. In addition, the investigators will collect provider and participant feedback at an exit interview immediately following the post-treatment assessment. The investigators will use multiple linear and logistic regression models to assess the effect of treatment on outcome measures across the study assessment time points.

ELIGIBILITY:
Inclusion Criteria:

* English speaking male and female Veterans ages 18-70;
* demonstrate an understanding of the informed consent;
* seeking or receiving services at the Canandaigua VA Medical Center (VAMC) or Rochester Outpatient Clinic;
* endorse death/suicidal ideation on the Columbia Suicide Severity Rating Scale
* either (i) a current diagnosis in their medical record of Major Depressive Disorder, Depression not otherwise specified, PTSD,or (ii) evidence of current depression as indicated by a score of > 10 on the Patient Health Questionnaire (PHQ-9) or current PTSD as indicated by a score of > 38 on the PTSD Symptom Checklist (PCL-5)();
* have an Insomnia Severity Index score > 10 indicating clinically meaningful insomnia with at least 1 insomnia-related daytime consequence (score of 1 on item #3) and trouble sleeping 3 months

Exclusion Criteria:

* history of serious mental illness such as schizophrenia, Bipolar I or II disorder, or current psychiatric conditions such as psychosis, mania, dementia, cognitive impairment, OR suicidal ideation with plan and intent, a report of a suicide attempt in the past 6 months in the Computerized Patient Record System (CPRS) or via self-report, or a score of 4 on the Columbia-Suicide Severity Rating Scale
* currently engaged in inpatient or partial hospitalization programs or ongoing/pending medical procedures that could inhibit sleep
* recent substance dependence disorder with < 3 months in remission or abstinence;
* suspicion of or evidence of untreated sleep apnea.
* Diagnosis of a circadian rhythm disorder
* Diagnosis of Narcolepsy
* History of Seizures

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2015-02; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wilfred R Pigeon, PhD, Principal Investigator — Syracuse VA Medical Center, Syracuse, NY
Locations (1):
- Syracuse VA Medical Center, Syracuse, NY, Syracuse, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 581 potential participants were identified from medical records and received a recruitment letter from their current treatment provider; 420 were reachable and screened by phone with 71 meeting initial eligibility criteria, completing written informed consent and baseline interview. 54 participants met all eligibility criteria and were randomized.
Groups:
- TAU Control: Treatment as Usual: All participants will be encouraged to begin or continue treatment of co-occurring conditions as recommended by treatment providers. This may include treatment within the primary care teams, through behavioral telehealth, and/or specialty outpatient mental health. Participants randomized to TAU may receive pharmacotherapy for insomnia, though CBT-I will be precluded until after the post-treatment assessments.
  TAU: Treatment as Usual: All participants will be encouraged to begin or continue treatment of co-occurring conditions as recommended by treatment providers. This may include treatment within the primary care teams, through behavioral telehealth, and/or specialty outpatient mental health. Participants randomized to TAU may receive pharmacotherapy for insomnia, though CBT-I will be precluded until after the post-treatment assessments.
Period: Overall Study
Arm/Group | CBT-I + TAU | TAU Control
Started | 26 | 28
Completed | 23 | 27
Not Completed | 3 | 1
Not completed — Lost to Follow-up | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CBT-I + TAU | TAU Control | Total
Number analyzed (Participants) | 26 | 28 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.9 (14.1) | 57.2 (10.8) | 55.4 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 20 | 23 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 25 | 27 | 52
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 4 | 9
  White | 17 | 21 | 38
  More than one race | 3 | 2 | 5
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 26 | 28 | 54

OUTCOME MEASURES:

1. Primary Outcome: Columbia Suicide Severity Rating Scale (C-SSRS)
Description: The entire Columbia Suicide Severity Rating Scale (C-SSRS) will be administered, but the investigators will use its' Suicidal Ideation Intensity scale (0-25 score range summed from five items, with higher scores indicating more severe suicidal ideation) as the primary outcome.
Time Frame: post-treatment (~6-8 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CBT-I + TAU | TAU Control
Number analyzed (Participants) | 23 | 27
units on a scale | 5.4 (6.8) | 8.4 (6.3)
Statistical Analysis 1: Comparison: CBT-I + TAU vs TAU Control; Test type: Superiority or Other; p = .153, Regression, Linear; multiple regression controlling for baseline values of the dependent variable was used to examine between group effects at post-treatment

2. Secondary Outcome: Perceived Treatment Beliefs (PTS)
Description: A 21-item measure (with items ranging from 1-7) based on the theory of planned behavior and designed to assess beliefs about treatment and plans to engage in treatment in military populations. This measure will focus on engagement in PTSD and depression treatments. The total score has a range of 21-147 with higher scores indicating higher likelihood of engaging in care.
Time Frame: post-treatment (~6-8 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CBT-I + TAU | TAU Control
Number analyzed (Participants) | 23 | 27
units on a scale | 135.7 (18.0) | 133.04 (28.8)
Statistical Analysis 1: Comparison: CBT-I + TAU vs TAU Control; Test type: Superiority or Other; p = .627, Regression, Linear

3. Secondary Outcome: Patient Health Questionnaire-9 (PHQ-9)
Description: A well-validated 9-item self-report measure developed to assess depression severity; higher scores are associated with greater severity (range of 0-27 with higher scores indicating more severe depression severity).
Time Frame: post-treatment (~6-8 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CBT-I + TAU | TAU Control
Number analyzed (Participants) | 23 | 27
units on a scale | 6.4 (4.6) | 12.3 (5.4)
Statistical Analysis 1: Comparison: CBT-I + TAU vs TAU Control; Test type: Superiority or Other; p < .001, Regression, Linear; [statistical method as in outcome 1, analysis 1]

4. Secondary Outcome: Insomnia Severity Index (ISI)
Description: A well-validated 7-item self-report measure developed to assess insomnia severity; higher scores are associated with greater severity (range of 0-28 with higher scores indicating greater insomnia severity).
Time Frame: post-treatment (~6-8 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CBT-I + TAU | TAU Control
Number analyzed (Participants) | 23 | 27
units on a scale | 7.9 (5.5) | 17.8 (5.2)
Statistical Analysis 1: Comparison: CBT-I + TAU vs TAU Control; Test type: Superiority or Other; p < .001, Regression, Linear; [statistical method as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: During study participation of approximately 8 weeks
Arm/Group | CBT-I + TAU | TAU Control
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/27
Other Adverse Events (participants affected / at risk) | 0/23 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No